CLINICAL TRIAL: NCT04206696
Title: Learning Curve for Minimally Invasive Oesophagectomy and Contrast With Open Procedure
Status: Completed | Type: Observational
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: MIE ZYP1
Record Dates: First submitted 2019-12-15; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Minimally Invasive Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Minimally invasive oesophagectomy is a technically demanding procedure; thus, the learning curve of this procedure should be explored. Then the mature minimally invasive oesophagectomy procedure should be contrasted with the open procedure.

DETAILED DESCRIPTION:
Between July 2010 and August 2016, 214 patients underwent MIE (thoracoscopic-laparoscopic oesophagectomy) for oesophageal squamous cell carcinoma in the Thoracic Department, The Second Hospital of Shandong University. Eight of these 214 patients were converted to thoracotomy or laparotomy, one patient was unable to tolerate single-lung ventilation due to a history of left upper lobectomy, and the other seven patients were due to bleeding controlling. Among the 214 patients enrolled, there were 182 males and 32 females in the MIE group. A total of 170 patients underwent oesophagectomy by open thoracotomy from August 2014 to August 2016, and these patients were defined as the open group. The data from the patients in the open group were compared with those of the patients who underwent thoracoscopic-laparoscopic oesophagectomy during the same clinical period. All patients were preoperatively diagnosed with oesophageal cancer by endoscopy and biopsy, with routine thoracic and abdominal enhanced computed tomography (CT) scans and endoscopic ultrasonography to evaluate the clinical TNM stage. The operations were performed by a single surgical team. This study was approved by the ethics committee and Medical Administration Division of the Second Hospital of Shandong University. Written informed consent was obtained from each of the enrolled patients. All methods performed in the investigator's study were conducted in accordance with the relevant guidelines and regulations.

ELIGIBILITY:
Inclusion Criteria:

oesophageal cancer diagnosed by endoscopy and biopsy good cardiopulmonary function to tolerate surgery

Exclusion Criteria:

poor cardiopulmonary function distant metastasis T4 with little possibility of radical resection

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were preoperatively diagnosed with oesophageal cancer by endoscopy and biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
bleeding volume | Between July 2010 and August 2016
  bleeding volume in milliliter
operation time | Between July 2010 and August 2016
  operation time in minutes
complications | Between July 2010 and August 2016
  complications in percentage
mortality | Between July 2010 and August 2016
  mortality in percentage
lymphadenectomy | Between July 2010 and August 2016
  lymphadenectomy in number

SECONDARY OUTCOMES:
2-year overall survival rate | Between August 2016 and August 2018
  2-year overall survival in percentage
2-year disease-free survival | Between August 2016 and August 2018
  2-year disease-free survival in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Xiaogang Zhao, Doctor, Study Director — The Second Hospital of Shandong University